CLINICAL TRIAL: NCT02029859
Title: Sleep Apnea, Obesity and Pregnancy
Acronym: GOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/070/HP
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Pregnancy
Keywords: pregnancy (after 30 weeks of amenorhea); obesity (BMI>35); sleep apnea syndrom; preeclampsy; intrauterine growth restriction
MeSH Terms: conditions — Obesity; Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prevalence of obstructive sleep apnea syndrome (Experimental): Determine the prevalence of obstructive sleep apnea syndrome (OSA) in late pregnancy in a population of obese patients .
  Polygraphic examination between 30 and 36 weeks of amenorhea
  Interventions: Procedure: Polygraphic examination

INTERVENTIONS:
Procedure: Polygraphic examination — Polygraphic examination between 30 and 36 weeks of amenorhea

SUMMARY:
Main objective:

Determine the prevalence of obstructive sleep apnea syndrome (OSA) in late pregnancy in a population of obese patients .

Secondary objectives :

* Identify risk factors for OSA during pregnancy (age, parity, high blood pressure, snoring , weight, neck circumference, scores on symptoms of sleep apnea, ... ) .
* Compare perinatal morbidity among obese patients with OSA in late pregnancy with case-controls.
* Evaluate the evolution of a moderate or severe OSA 6 months after pregnancy.

Material and methods

Characteristics of the study:

* Interventional biomedical research
* Prospective Multicenter nonrandomized study

Flow chart

* Patients will be included between 30 and 36 weeks of amenorrhea (WA) .
* Will rated from inclusion: age, parity, weight, height, BMI in early pregnancy, neck circumferrence, treated high blood pressure.
* As recommended in France, the main test results during the pregnancy follow-up will be recorded.
* At the inclusion visit will be conducted a Berlin Questionnaire and Epworth Score.
* Screening for OSA by nocturnal polysomnography will be performed between 30 and 36WA. This screening can be performed as an outpatient.
* In case of proven OSA patients will be offered an appropriate care by today's standards.
* Whatever the outcome of pregnancy, a second polysomnography will be performed 6 months after childbirth in case of OSA during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* BMI >35
* Pregnancy after 30 Weeks of amenorhea
* Age > 18
* Signed consentment
* Nationnal Health Program affiliation

Exclusion Criteria:

* Twin or more pregnancy
* Imprecise term
* Artificial insemination with donor gametes
* Proved thrombophilia
* chronic renal failure
* Previously treated (with CPAP) obstructive sleep apnea syndrom

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sleep apnea syndrom prevalence | 6 weeks
  Polygraphic examination for all subjects will determine the sleep apnea syndrom prevalence during late pregnancy (after 30 weeks of amenorhea) for severe obese women (BMI>35).

CONTACTS AND LOCATIONS:
Overall Officials: Loic Marpeau, PHD, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - Angers University Hospital, Angers
  - Caen University Hospital, Caen
  - Le Havre Hospital, Le Havre
  - Rouen University Hospital, Rouen